CLINICAL TRIAL: NCT02439567
Title: Usefulness of Transient Elastography Assessing Liver Fibrosis and Portal Hypertension in Patients With HCV Cirrhosis Treated With New All Oral Antiviral Drugs
Brief Title: Transient Elastography to Assess Liver Fibrosis and Portal Hypertension in HCV Cirrhotic Patients Treated With New Antiviral Drugs (SPLEEN-C)
Acronym: SPLEEN-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SPLEEN-C (JOA-SOF-2015-01)
Record Dates: First submitted 2015-04-27; First posted 2015-05-08 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Chronic Hepatitis C; Cirrhosis; Portal Hypertension
Keywords: Cirrhosis; Chronic hepatitis C; Clinically significant portal hypertension; Portal hypertension; Elastography; Antiviral therapy
MeSH Terms: conditions — Hepatitis C, Chronic; Fibrosis; Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Experimental): Treatment with new oral antiviral drugs for HCV infection, Fibroscan: Liver and Spleen elastography
  Interventions: Device: Fibroscan: Liver and Spleen elastography

INTERVENTIONS:
Device: Fibroscan: Liver and Spleen elastography — In cirrhotic patients treated with antivirals for HCV infection, repeated liver and spleen stiffness measures with Fibroscan will be performed to predict the presence of clinically significant and severe portal hypertension.

SUMMARY:
The purpose of this study is to evaluate the effects of sustained virological response in liver and spleen stiffness in patients with HCV compensated advanced chronic liver disease treated with new all oral antiviral drugs in order to determine factors implicated in stiffness change and its implications for long-term follow-up.

DETAILED DESCRIPTION:
Prospective cohort study including consecutive patients (with baseline liver stiffness measurement ≥10 kPa who meet the Baveno VI criteria for compensated advanced chronic liver disease) who initiate treatment with new all oral antiviral drugs following current recommendations in Spain.

In all these patients the following parameters will be assessed:

* Baseline liver and spleen stiffness and CAP measurements at the time of starting therapy and then, during treatment in week 4 and week 12 (end of treatment). After finishing therapy, these measurements will be repeated at 6 and 12 months of follow-up.
* Routine lab tests, including liver enzymes and viral load, will be performed at baseline, 4 and 12 weeks of therapy, and at 3 and 6 months after finishing therapy according to standard clinical practice.
* Liver ultrasound will be performed every 6 months as a routine procedure in patients wiht liver cirrhosis.
* Patients who were known to have esophageal varices prior to therapy will be assessed with an upper endoscopy 12 months after finishing therapy if they achieve SVR.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 90 years.
* History of chronic hepatitis C infection.
* Compensated advanced chronic liver disease (Baveno VI definition):

  * Baseline liver stiffness ≥15 kPa or,
  * Baseline liver stiffness 10-15 kPa and one of the following: platelet count <150x10e9/L, spleen size ≥13 cm, nodular liver or collateral circulation in abdominal ultrasound, HVPG >5 mmHg, upper gastrointestinal endoscopy showing gastroesophageal varices or previous liver biopsy showing bridging fibrosis or cirrhosis.
* Indication to start antiviral treatment with new oral drugs.
* Willingness to enter the study.
* Sign the informed consent.

Exclusion Criteria:

* Chronic liver disease due to other etiology than HCV.
* Terminal illness.
* Treatment with interferon.
* Liver stiffness measurement < 10 kPa at baseline.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Liver stiffness change during treatment and at 6 months of follow-up in patients who achieve sustained virological response (SVR). | 6 months
Spleen stiffness change during treatment and at 6 months of follow-up in patients who achieve SVR. | 6 months

SECONDARY OUTCOMES:
Overall survival (Composite outcome including survival free of all cause of death, liver transplantation, decompensation and/or increase in >1 point in Child Pugh score). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Joan Genescà Ferrer, PhD MD, Principal Investigator — Hospital Universitari Vall d'hebron Barcelona, Spain
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain